CLINICAL TRIAL: NCT00726895
Title: A Randomized, Two-way Crossover Design Used to Compare the Dose Proportionality of Quinine Sulfate Capsules, 324 mg Following a Single Oral Dose of 1 x 324 mg Capsule Versus 2 x 324 mg Capsules in Healthy Adult Volunteers
Brief Title: A Dose Proportionality Study of Quinine Sulfate Capsules Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Matthew W. Davis, MD,, Mutual Pharmaceutical
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: R04-0376
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2009-12-30 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Bioavailability
MeSH Terms: interventions — Quinine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quinine Sulfate Capsules 1 x 324 mg Dose (Experimental): Quinine Sulfate 1 x 324 mg capsule dose.
  Interventions: Drug: Quinine Sulfate Capsules 324 mg
- Quinine Sulfate Capsules 2 x 324 mg Dose (Experimental): Quinine Sulfate 2 x 324 mg capsules dose.
  Interventions: Drug: Quinine Sulfate Capsules 324 mg

INTERVENTIONS:
Drug: Quinine Sulfate Capsules 324 mg — 1 x 324 mg capsule
  Arms: Quinine Sulfate Capsules 1 x 324 mg Dose
Drug: Quinine Sulfate Capsules 324 mg — 2 x 324 mg capsules
  Arms: Quinine Sulfate Capsules 2 x 324 mg Dose

SUMMARY:
The purpose of this study is to evaluate and compare the dose proportionality of 324 mg Quinine Sulfate capsules following a single oral dose (1 x 324 mg capsules versus 2 x 324 mg capsules) in healthy adult volunteers when administered under fasting conditions.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and compare the dose proportionality of 324 mg Quinine Sulfate capsules following a single oral dose (1 x 324 mg capsules versus 2 x 324 mg capsules) in healthy adult volunteers when administered under fasting conditions.

Twenty-four healthy, non-smoking, non-obese, male and female volunteers at least 18 years of age will be randomly assigned in a crossover fashion to receive each of two Quinine Sulfate dosing regimens in sequence with a 7 day washout period between dosing periods. On the morning of Day 1, after an overnight fast of at least 10 hours, subjects will receive either a single oral dose of treatment A, Quinine Sulfate 1 x 324 mg capsule, or a single oral dose of treatment B, Quinine Sulfate 2 x 324 mg capsules. After a 7 day washout period,on the morning of Day 8 following an overnight fast of at least 10 hours, subjects will receive the alternate regimen. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of Quinine Sulfate. Blood sampling will then continue on a non-confined basis at 36 and 48 hours post-dose. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout the confinement portion of the study for adverse reactions to the study drug and/or procedures. Blood pressure and heart rate will be obtained prior to dosing and as scheduled following each dose. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All volunteers will be healthy men or women 18 years of age or older at the time of dosing. The weight range will not exceed ±20% for height and body frame as per Desirable Weights for Adults - 1983 Metropolitan Height and Weight Table
* Screening procedures: Each volunteer will complete the screening process within 28 days prior to Period I dosing. Consent documents for both screening evaluation and human immunodeficiency virus (HIV) antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures
* Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.
* The screening clinical laboratory procedures will include:
* HEMATOLOGY: hematocrit, hemoglobin, white blood cell (WBC) count with differential, red blood cell (RBC) count, platelet count;
* CLINICAL CHEMISTRY: serum creatinine, blood urea nitrogen (BUN), glucose, AST(SGOT - Serum glutamic-oxaloacetic transaminase), ALT(SGPT - Serum glutamic-pyruvic transaminase), albumin, total bilirubin, total protein, and alkaline phosphatase;
* HIV antibody and hepatitis B surface antigen screens;
* URINALYSIS: by dipstick; full microscopic examination if dipstick positive; and
* URINE DRUG SCREEN: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine
* SERUM PREGNANCY SCREEN (female volunteers only)

If female and:

* of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condom with spermicide, diaphragm, intrauterine device (IUD), or abstinence; or
* is postmenopausal for at least 1 year; or is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators)
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant
* Volunteers demonstrating a positive hepatitis B surface antigen screen or a reactive HIV antibody screen
* Volunteers demonstrating a positive drug abuse screen when screened for this study
* Female volunteers demonstrating a positive pregnancy screen
* Female volunteers who are currently breastfeeding
* Volunteers with a history of allergic response(s) to quinine or related drugs
* Volunteers with a history of clinically significant allergies including drug allergies
* Volunteers with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators)
* Volunteers who currently use tobacco products
* Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing
* Volunteers who report donating greater than 150 mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study
* Volunteers who have donated plasma (e.g.plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study
* Volunteers who report receiving any investigational drug within 28 days prior to Period I dosing
* Volunteers who report taking any systemic prescription medication in the 14 days prior to Period I dosing
* Volunteers with a QTc (corrected QT interval) > 480 msec on the screening electrocardiogram (ECG) or with clinically significant findings
* Volunteers who have a glucose-6-phosphate dehydrogenese deficiency (G6PD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-05; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Quinine Sulfate Capsules 1 x 324 mg Dose Then 2 x 324 mg Dose; Quinine Sulfate Capsules 2 x 324 mg Dose Then 1 x 324 mg Dose: All subjects received each of the two study regimens (Treatment A - Quinine Sulfate 1 x 324 mg capsule, Treatment B - Quinine Sulfate 2 x 324 mg capsules) in a randomly assigned sequence of dosing periods, each followed by a washout period of 7 days.
Period: First Intervention
Arm/Group | Quinine Sulfate Capsules 1 x 324 mg Dose Then 2 x 324 mg Dose | Quinine Sulfate Capsules 2 x 324 mg Dose Then 1 x 324 mg Dose
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Quinine Sulfate Capsules 1 x 324 mg Dose Then 2 x 324 mg Dose | Quinine Sulfate Capsules 2 x 324 mg Dose Then 1 x 324 mg Dose
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Quinine Sulfate Capsules 1 x 324 mg Dose Then 2 x 324 mg Dose | Quinine Sulfate Capsules 2 x 324 mg Dose Then 1 x 324 mg Dose
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received either one Quinine Sulfate 324 mg capsule or two Quinine Sulfate 324 mg capsules following an overnight fast of at least 10 hours.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma.
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36 and 48 hours after drug administration.
Population: Plasma concentration data for 23 of the 24 enrolled subjects were used in the statistical analysis. Subject number 12 dropped from the study prior to period II (Treatment A) dosing. Treatment A, Dose Adjusted to 2 x 324 mg was a statistical adjustment only used to evaluate for dose proportionality.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Treatment A - Quinine Sulfate Capsules (1 x 324 mg Dose): Each subject received one capsule of Quinine Sulfate 324 mg after an overnight fast of at least 10 hours.
- Treatment A, Dose Adjusted to 2 x 324 mg: This group was a statistical adjustment only. Treatment A (Quinine Sulfate 1 x 324 mg Capsule) Dose Adjusted to 2 x 324 mg was used to evaluate for dose proportionality.
- Treatment B - Quinine Sulfate Capsules (2 x 324 mg Dose): Each subject received two capsules of Quinine Sulfate 324 mg after an overnight fast of at least 10 hours.
Arm/Group | Treatment A - Quinine Sulfate Capsules (1 x 324 mg Dose) | Treatment A, Dose Adjusted to 2 x 324 mg | Treatment B - Quinine Sulfate Capsules (2 x 324 mg Dose)
Number analyzed (Participants) | 23 | 23 | 23
ng/mL | 2,118.35 (517.79) | 4,236.70 (1,035.58) | 3,242.92 (685.80)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Treatment A - Quinine Sulfate Capsules (1 x 324 mg Dose) | Treatment A, Dose Adjusted to 2 x 324 mg | Treatment B - Quinine Sulfate Capsules (2 x 324 mg Dose)
Number analyzed (Participants) | 23 | 23 | 23
ng-hr/mL | 31,951.03 (10,428.59) | 63,902.06 (20,857.17) | 56,198.20 (15,683.25)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Treatment A - Quinine Sulfate Capsules (1 x 324 mg Dose) | Treatment A, Dose Adjusted to 2 x 324 mg | Treatment B - Quinine Sulfate Capsules (2 x 324 mg Dose)
Number analyzed (Participants) | 23 | 23 | 23
ng-hr/mL | 35,199.28 (12,678.60) | 70,398.56 (25,357.19) | 61,570.10 (19,295.34)

ADVERSE EVENTS:
Description: 24 subjects were enrolled in this study. One subject dropped out of the study prior to receiving both interventions. 23 subjects were administered the Quinine Sulfate 1 x 324 mg capsule dose and 24 subjects were admistered the Quinine Sulfate 2 x 324 mg capusle dose.
Groups:
- Treatment A - Quinine Sulfate Capsules 1 x 324 mg Dose; Treatment B - Quinine Sulfate Capsules 2 x 324 mg Dose: All subjects received each of the two study regimens (Treatment A - Quinine Sulfate 1 x 324 mg capsule, Treatment B - Quinine Sulfate 2 x 324 mg capsules) in a randomly assigned sequence of dosing periods, each followed by a washout period of 7 days.
Arm/Group | Treatment A - Quinine Sulfate Capsules 1 x 324 mg Dose | Treatment B - Quinine Sulfate Capsules 2 x 324 mg Dose
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 6/23 | 10/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A - Quinine Sulfate Capsules 1 x 324 mg Dose (N=23) | Treatment B - Quinine Sulfate Capsules 2 x 324 mg Dose (N=24)
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Generalized pain (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Joint injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia in extremities (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (General disorders) | 0 (0) | 1 (1)
Pallor (General disorders) | 1 (1) | 1 (1)
Pharyngolaryngeal - Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rigors (General disorders) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sweating increased (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Tinnitus (Nervous system disorders) | 0 (0) | 1 (1)
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days